CLINICAL TRIAL: NCT06343012
Title: Effect of Caring Leadership Intervention Program for First-Line Nurse Managers on Their Managerial Actions and Nurse Outcomes
Brief Title: Caring Leadership Intervention Program for First-Line Nurse Managers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matrouh University (Other)
Responsible Party: Principal Investigator, Nagah Abd El-Fattah Mohamed Aly, Assistant professor of Nursing administration, Matrouh University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 0305900
Record Dates: First submitted 2024-03-27; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Intervention; Behavior
Keywords: Caring; Leadership; Management; Actions; Nurse; Outcmes
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: A quasi-experimental study design utilized two groups, study and control groups
Who Masked: Participant
Masking Description: A quasi-experimental study design utilized two groups, study and control groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): The study group received the Caring Leadership Intervention program
  Interventions: Other: Caring leadership Intervention program
- Control group (Other): The control group did not receive the caring leadership intervention program
  Interventions: Other: Caring leadership Intervention program

INTERVENTIONS:
Other: Caring leadership Intervention program — Caring leadership intervention program

SUMMARY:
Caring leadership can help first-line nurse managers create a healthy environment, resulting in a positive outcome for nurse staff, patients, and healthcare organizations.

DETAILED DESCRIPTION:
Developing caring behaviors among nurse managers is critical for establishing an effective nursing care environment. Enhancing the caring leadership of nurse managers would lead to improving nurses' perception regarding nurse manager caring behaviors and positive nurse outcomes. This study aimed to Examine the effect of a caring leadership intervention program for first-line nurse managers on their caring knowledge and managerial actions as well as nurses' perceived first-line nurse managers' nurse outcomes..

ELIGIBILITY:
Inclusion Criteria:

First nurse managers

* Work in inpatient wards and intensive care units
* Sign the informed consent

Exclusion Criteria:

First nurse managers

* Refuse to provide consent
* Decline to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Questionnaire to measure first-line nurse managers' knowledge | one month
  Knowledge of 60 first-line nurse managers as assessed using a binary scale (0= No, 1= Yes). Change in nurse managers' knowledge level in three months.
Questionnaire to measure the managerial actions of first-line nurse managers | Two months
  First-line nurse manager actions as assessed by a five- Likert scale (From 1 (never) to 5 (always)).
  Change in nurse manager actions in two months.
Questionnaire to assess nurses' perceived first-line nurse managers' caring behavior | one month
  Nurses' perceived first-line nurse managers' caring behavior as assessed by a 5-point Likert-type scale from 1 (never) to 5 (always). Change of nurses' perception in one month.
questionnaire to measure nurse outcomes | two months
  nurse outcomes (job satisfaction and work engagement)as assessed by a five- Likert scale.Change in nurse outcomes in two months

CONTACTS AND LOCATIONS:
Overall Officials: Nagah Abd El-Fattah Mohamed Aly, Ph.D, Study Chair — Faculty of Nursing, Matrouh University, Egypt; Wael M. Lotfy, Ph.D, Study Director — Faculty of Nursing, Matrouh University, Egypt
Locations (1):
- Faculty of Nursing, Matrouh University, Marsá Maţrūḩ, Egypt

IPD SHARING:
Plan to Share IPD: No